CLINICAL TRIAL: NCT03526276
Title: Effect of Fluoride and Casein Phosphopeptide-amorphous Calcium Phosphate on Remineralization of Early Caries Lesions in Primary Teeth: an in Vivo Study
Brief Title: Effect of Different Pastes on Remineralization of Early Caries Lesions in Primary Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Collaborators: Scientific Research Fund, Ministry of Higher Education and Research, Jordan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 284-2015
Record Dates: First submitted 2017-03-06; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2017-03

CONDITIONS: White Spot Lesion of Tooth
Keywords: Quantitative Laser Fluorescence (QLF); CPP-ACP paste; Fluoride toothpaste; Combined use of fluoride and CPP-ACP paste; Primary teeth
MeSH Terms: interventions — Fluorides; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial involving 118 children ages between 4 and 5 years. They will be examined and chosen randomly for the study. Children will be divided equally into three groups: Group 1 will use CPP-ACP twice daily, Group 2 will apply fluoridated toothpaste twice daily, Group 3 will apply fluoridated toothpaste and CPP-ACP twice daily. Quantitative assessment of white spot lesions will be carried out using QLF before remineralizing agent application (baseline) and at 3, and 6 month intervals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CPP-ACP paste (Active Comparator): Casein phosphopeptide amorphous calcium phosphate is a product that contains calcium, phosphate, protein and casein.
  Interventions: Other: CPP-ACP paste
- Fluoride toothpaste (Active Comparator): Fluoride toothpaste
  Interventions: Other: Fluoride toothpaste
- Both (Fluoride and CPP-ACP) (Active Comparator): Fluoride toothpaste and CPP-ACP paste
  Interventions: Other: Both (Fluoride and CPP-ACP)

INTERVENTIONS:
Other: CPP-ACP paste — Children will brush their teeth with CPP-ACP paste twice daily.
  Arms: CPP-ACP paste
Other: Fluoride toothpaste — Children will brush their teeth with fluoridated toothpaste twice daily
  Arms: Fluoride toothpaste
Other: Both (Fluoride and CPP-ACP) — Children will brush their teeth with fluoridated toothpaste and apply CPP-ACP immediately after toothbrushing, twice daily.
  Arms: Both (Fluoride and CPP-ACP)

SUMMARY:
This study is a randomized controlled trial involving 118 children ages between 4 and 5 years to assess the remineralization effect of Casein Phosphopeptide-Amorphous Calcium Phosphate (CPP-ACP) on white spot lesions in primary teeth using Quantitative Light-induced Fluorescence (QLF) system, and compare that with fluoride alone or combined use of fluoride and CPP-ACP.

DETAILED DESCRIPTION:
Aim: To assess the remineralization effect of CPP-ACP on white spot lesions in primary teeth using QLF system, and compare that with fluoride alone or combined use of fluoride and CPP-ACP.

Materials and Methods:

o Study design:

The present study is a randomized control trial (RCT).

* Study setting: The present study will be conducted at Kindergartens, Irbid, Jordan. A list of schools will be obtained from the development sector, schools will be invited to be participate in the study. Children will be randomly allocated into groups.
* Study procedure:

  * Study population includes healthy children (n=118) aged between 4-5 years diagnosed with white spot lesions.
  * Oral examination at baseline to record dmft and caries risk using the Caries-risk Assessment Tool (CAT) based on American Academy of Pediatric Dentistry (AAPD) guidelines will be carried out, patients will be classified as: low, moderate or high risk
  * Quantitative assessment of early caries lesions will be carried out using QLF.
  * Children will be randomly allocated into three groups:

Group 1: children will brush their teeth with CPP-ACP twice daily.

Group 2: children will brush their teeth with fluoridated toothpaste twice daily.

Group 3: children will brush their teeth with fluoridated toothpaste and apply CPP-ACP immediately after tooth brushing, twice daily.

The researcher will do the morning application at school, the evening application will be done at home with help of the parent. The researcher will give oral hygiene and brushing instructions to the parents and also diet advice. An oral hygiene chart will be given to monitor twice-daily tooth brushing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 4-5 years old children, with primary dentition, and early white spot lesions

Exclusion Criteria:

* Lack of cooperation in the oral examination.
* Allergies to milk protein.
* Have received a fluoride supplement or professional topical fluoride application at least 3 months before or during the study period.
* Medically compromised patient.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change in remineralization of white spot lesions using Quantitative Light-induced Fluorescence (QLF) machine | 3 and 6 months
  Change in remineralization of white spot lesions as indicated by changes in fluorescence levels detected by QLF after use of CPP-ACP, Fluoride or both agents over 3 and 6 months.

SECONDARY OUTCOMES:
Changes in caries using the decayed, missing due to caries, filled, deciduous teeth (dmft) index. | 3 and 6 months
  Changes in dmft after use of CPP-ACP, Fluoride or both agents over 3 and 6 months.
Changes in caries using the decayed, missing due to caries, filled, deciduous tooth surfaces (dmfs) index. | 3 and 6 months
  Changes in dmfs after use of CPP-ACP, Fluoride or both agents over 3 and 6 months.
Changes in caries using the International Caries Detection and Assessment System (ICDAS) scores. | 3 and 6 months
  Changes in ICDAS scores over 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Al-Batayneh, MDSc, FRACDS, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No